CLINICAL TRIAL: NCT03991598
Title: Connecting Emergency Departments With Community Services to Prevent Mobility Losses in Pre-frail & Frail Seniors (CEDeComS)
Brief Title: Connecting Emergency Departments With Community Services to Prevent Mobility Losses in Pre-frail & Frail Seniors
Acronym: CEDeComS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Université du Québec a Montréal (Other); University of Toronto (Other); Laval University (Other); Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other); Ottawa Hospital Research Institute (Other); Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other); Alberta Health Services, Calgary (Other); Sunnybrook Research Institute (Other); Washington University School of Medicine (Other); McMaster University (Other); Mount Sinai Hospital, Canada (Other); The Ottawa Hospital (Other); Université de Montréal (Other); University of Ottawa (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Marie-Josée Sirois, Ph.D Independent Researcher - Mid Career Investigator, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MP-20-2017-3235; 364485 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2017-07-19; First posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Elderly; Functional Status
Keywords: Frail; Prefrail; Mobile decline
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: This is a step-wedge clinical trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): EDs 1 to 7 will then be randomly phased-in INT every 3 months.
  Interventions: Other: Exercise program
- control (No Intervention): During the first 6 months and throughout CTRL time

INTERVENTIONS:
Other: Exercise program — Exercise program in communities / Exercise program at home
  Arms: intervention

SUMMARY:
About 18% of independent people over 65 who are evaluated in Emergency Departments for minor injuries (fractures, sprains) present some mobility decline up to 3 to 6 months postinjury. People at risk of decline are prefrail or frail; this condition could be explained by muscle proprieties loss. Exercise is a proven method that can help limit frailty and allow to restore mobility.

The aim of our study is to evaluate whether a suitable exercise program of one hour, twice a week for 12 weeks will limit functional losses & fragility in injured older adults after their emergency department visit.

DETAILED DESCRIPTION:
Yearly, around 400 000 Canadian community-dwelling seniors sustain injuries that are not life threatening but limit their mobility and normal activities. Up to 65 % of these seniors seek care in Emergency Departments (EDs) and 2/3 are discharged from EDs with varying degrees of minor injuries. Since 2010 and using multicenter large Canadian cohorts (n=3000), our CIHR CETI* emerging team has shown that minor injuries trigger a downward spiral of mobility decline in 16% of seniors who are still independent at the time of injury, unmasking early impairments and a prefrail or frail status. As there are no ED management guidelines designed to prevent these prefrail (35%) and frail (13%) injured seniors from losing their mobility and function, they do deteriorate within 6 months post-ED discharge. This is unfortunate because there is compelling evidence of the effectiveness of community and home-based mobility interventions showing that simple, targeted interventions can prevent frailty and functional limitations.

In that context, identification of seniors at risk in EDs is crucial to implement effective interventions. The CETI has validated a simple Clinical Decision Rule (CETI-CDR) that screens and orients seniors at high, moderate and low risk of functional decline to appropriate post-ED follow-ups. The latter include effective community-based mobility interventions available across all Canadian communities. An ongoing pilot study (n=120) in two EDs is showing the feasibility and effectiveness (functional decline prevention) of interventions and patient satisfaction. The investigators thus propose to implement the CEDeComS intervention, which involves the CETI-CDR combined with rapid linkage to community mobility programs directly from EDs.

The Main Objectives of this study are to 1) evaluate the effectiveness of the CEDeComS compared to usual care, on improving seniors' health outcomes, 2) determine the cost-effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Consultation at Emergency Department (ED) for an injury
* Injury happened in the 14 days prior to ED visit
* 65 years old and over
* Discharge from ED within 48 hours
* Independant in basic Activities of Daily Living (ADL)

Exclusion Criteria:

* Hospitalization related to the trauma
* Major surgery related to the trauma
* Not independant in ADL
* Living in a long-term care home
* Important cognitive impairment
* Not speaking French or English
* Unable to consent
* No trauma

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Changes in Cumulative Incidence of Functional Decline at 3 and 6 months after the intial ED visit (Baseline) | Outcome measures are assessed at three time points : Baseline T0: time of the Emergency Department (ED) consultation by participants T1: 3 months post-ED consultation; T2: 6 months post-ED consultation
  Proportions of participants showing, at 3 or 6 months post-ED visit, a loss ≥2/28 on the OARS scale, compared to Baseline. (OARS: Older American Resource and Services multidimensional functional scale, which includes 7 basic ADLs and 7 instrumental ADLs items)

SECONDARY OUTCOMES:
Changes in mean SPPB scores at 3 and 6 months after the initial ED visit (baseline) | Outcome measures are assessed at three time points : Baseline T0: time of the Emergency Department (ED) consultation by participants T1: 3 months post-ED consultation; T2: 6 months post-ED consultation
  The SPPB (Short Physical Portable Battery) combines walking, balance and strength items. Scores range from 0 to 12 (best).
Changes in mean SOF Frailty index scores at 3 and 6 months after the initial ED visit (from Baseline) | Outcome measures are assessed at three time points : Baseline T0: time of the Emergency Department (ED) consultation by participants T1: 3 months post-ED consultation; T2: 6 months post-ED consultation
  The SOF index is a Frailty measure. Scores range from 0/3 (robust senior) to 3/3 (frail senior)

CONTACTS AND LOCATIONS:
Overall Officials: Marcel ME Emond, Md, Ph.D, Principal Investigator — Centre de recherche du CHU de Québec
Locations (6):
- Canada (6):
  - Alberta Health Services, Calgary, Alberta
  - Alberta Health Services, Edmonton, Alberta
  - Sunnybrook Health Science Center, Toronto, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontaro
  - Hôpital Sacré-Coeur, Montreal, Quebec
  - CHU-Québec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Sirois MJ, Blais J, Aubertin-Leheudre M, Carmichael PH, Fruteau de Laclos L, Desjardins A, Daoust R, Eagles D, Lee J, Perry JJ, Salbach NM, Emond M. Effectiveness of Exercise in Older Adults Discharged From the ER After Minor Injuries: The CEDeComS Stepped-Wedge Trial. J Am Geriatr Soc. 2026 Jan;74(1):74-84. doi: 10.1111/jgs.70166. Epub 2025 Oct 20. PMID 41116303
- [Derived] Sirois MJ, Carmichael PH, Daoust R, Eagles D, Griffith L, Lang E, Lee J, Perry JJ, Veillette N, Emond M; Canadian Emergency Team Initiative on Mobility in Aging. Functional Decline After Nonhospitalized Injuries in Older Patients: Results From the Canadian Emergency Team Initiative Cohort in Elders. Ann Emerg Med. 2022 Aug;80(2):154-164. doi: 10.1016/j.annemergmed.2022.01.041. Epub 2022 Mar 16. PMID 35305850